CLINICAL TRIAL: NCT06949436
Title: Ultra-early Gamma Knife Stereotactic Radiosurgery for Trigeminal Neuralgia: Feasibility and Potential Benefit
Brief Title: Ultra-Early Gamma Knife Stereotactic Radiosurgery for TN
Acronym: URGEnt-TN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRS-0301
Record Dates: First submitted 2025-04-10; First posted 2025-04-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Trigeminal Neuralgia (TN)
Keywords: trigeminal neuralgia; Gamma Knife; stereotactic radiosurgery; surgery
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Intervention Model Description: Investigators will perform a single-centre, two-arm, randomized, controlled, parallel group design, pragmatic, noninferiority, phase II trial of ultra-early GK-SRS for trigeminal neuralgia in patients treated prior to developing a medically-refractory state and within 2 years of disease onset.
  Two parallel cohorts will be studied independently of each other: patients treated with GK-SRS (surgical arm/treatment group) versus pre-refractory patients treated with ongoing best medical management (medical arm/control group). Crossover will be allowed from the medical arm to the surgical arm. An intention-to-treat analysis will be carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (No Intervention): Patients allocated to the standard arm will continue their medical management per the judgment of treating physician.
- Gamma Knife stereotactic radiosurgery for TN (Experimental)
  Interventions: Procedure: GK SRS

INTERVENTIONS:
Procedure: GK SRS — Under local anaesthesia, a Leksell stereotactic head frame is fixed to the patient's head to allow for complete cranial immobilization during treatment. The retrogasserian (i.e., mid-cisternal) target will be utilized at a single 4 mm isocenter, and 40 Gy will be administered to the 50% isodose line while limiting the brainstem to 12 Gy.
  Arms: Gamma Knife stereotactic radiosurgery for TN

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and potential benefit of Gamma Knife stereotactic radiosurgery (GK-SRS) as an ultra-early treatment option for trigeminal neuralgia (TN).

The main questions it aims to answer are:

1. will earlier GK-SRS provide more durable pain relief compared to later GK-SRS?
2. will earlier GK-SRS reduce or eliminate the need for high-dose medical therapy?
3. will earlier GK-SRS have a lower risk of serious complications compared to other first-line treatments?

If participants are assigned to GK-SRS treatment group, they will be asked to:

• Undergo a preoperative MRI, measurements of heart rate and blood pressure, stereotactic head-frame placement, post-operative management and observation.

Both groups will be asked to:

* Complete medical histories and neurological examinations. These are part of standard of care.
* Participants will be asked a series of questions related to overall physical health, pain severity, and mood. Completing these questionnaires is part of the research activity. It will take approximately 15- 30 minutes to complete. These questionnaires include: The Barrow Neurological Institute Pain Intensity Score, Brief Pain Inventory-Facial (BPI-Facial), Visual Analog Scale (VAS), Medication Quantification Scale (MQS), Hospital Anxiety and Depression Scale (HADS), Pain Catastrophizing Scale (PCS), and the Short Form Health Survey.

DETAILED DESCRIPTION:
Background Trigeminal neuralgia (TN) is a chronic, often debilitating, neuropathic facial pain condition with an approximate global incidence of 12 cases per 100,000 and a female predominance of 3:2, occurring predominantly in the sixth decade of life and increases with age, peaking around 70 years. According to the International Classification of Headache Disorders (ICHD-3), TN is characterized by "recurrent unilateral brief electric shock-like pains, abrupt in onset and termination, limited to the distribution of one or more divisions of the trigeminal nerve (cranial nerve five - CNV) and triggered by innocuous stimuli". The CNV divides into three distinct subdivisions that carry sensory information from the scalp, forehead, eyes, upper and lower eyelids, mucous membranes of the nasal and oral cavities, frontal sinus, cheeks, teeth, lower and upper lips, and deep structures within the head. The severe lancinating pain of TN may be triggered by common somatosensory stimuli experienced in everyday life, such as chewing, speaking, brushing teeth, temperature changes, or tactile pressure to the face; pain attacks may also occur entirely spontaneously.

Given the severity of this condition, prompt pain management is critically important. Generally, pharmaceutical therapy is employed as the first-line treatment, usually in the form of antiepileptic drugs which are known to be effective against neuropathic pain, with carbamazepine (CBZ) being the gold standard. Unfortunately, these agents pose a significant risk of adverse effects ranging from ataxia, double vision, hyponatremia, confusion, and tremor, to more severe complications such as cardiac arrhythmia, aplastic anemia, hepatotoxicity, toxic epidermal necrolysis, and dosages reaching toxic levels. Frequently, increased doses are required to maintain therapeutic pain relief over time. Indeed, while pharmaceuticals may be the standard first-line treatment for TN, >50% of patients eventually fail medical therapy. The combination of unfavourable adverse effects and diminished drug response can lead to prolonged disruption of overall well-being in a considerable proportion of patients with TN.

In general, surgical options (i.e., microvascular decompression (MVD), percutaneous rhizotomy (PR), and Gamma Knife stereotactic radiosurgery (GK-SRS)) are reserved for patients who are classified as "medically refractory". In essence, surgical treatment is offered as a rescue therapy when pharmaceutical management has failed. Of the surgical options, GK-SRS is a highly precise type of radiation therapy which is by far the least invasive, carrying with it the lowest risk of serious adverse surgery-related risks. There is good evidence to support the safety and efficacy of GK-SRS in medically-refractory TN, with some data suggesting that earlier intervention (within 3-4 years of pain onset) may result in better long-term pain outcomes. However, what is not known is whether ultra-early intervention with GK-SRS-before the actual development of medical-refractoriness-could somehow alter the natural progression of TN, thereby avoiding the need for high-dose medical therapy altogether and the side effects associated with it.

Objective

The investigators aim to evaluate the feasibility and potential benefit of GK-SRS as an ultra-early treatment option for TN. Given the well-established tolerability of GK-SRS, it is hypothesized that ultra-early GK-SRS will:

1. provide more durable pain relief compared to later GK-SRS;
2. reduce or eliminate the need for high-dose medical therapy; and
3. have a lower risk of serious complications compared to other first-line treatments.

Treatment Given the overlap between the pain of TN and other craniofacial pain entities, treatment is often delayed due to misdiagnosis. Indeed, TN patients frequently undergo unnecessary dental procedures, given the predominant localization of symptoms within the maxillary and mandibular facial dermatomes, before a correct diagnosis is made. In addition, patients presenting to primary care or emergency medical physicians with persistent and debilitating pain may be erroneously prescribed analgesics-such as opioids-which are ineffective in suppressing neuropathic TN pain.

Early recognition of TN is imperative in mitigating prolonged suffering and the potentially disabling repercussions of untreated pain. It has been shown that duration of disease may play an important role in treatment refractoriness, which argues in favour of early intervention. As mentioned above, typically medical therapy with pharmacological agents is trialled as the initial pain management strategy; in the case of intolerability or the development of medical refractoriness, surgical options are then explored as the next step.

Medical Therapy Carbamazepine and Oxcarbazepine The general recommendation for first-line TN treatment is a trial of carbamazepine (CBZ), an antiepileptic medication used for its analgesic properties. CBZ specifically targets voltage-gated sodium channels by altering sodium availability during synaptic impulses, reducing or inhibiting neuronal excitability, which serves to reduce repetitive neuropathic pain signalling.

In its earliest clinical utilization for TN, CBZ produced promising results in a small cohort of patients. A subsequent study conducted by Blom, reported that 90% of patients had a favourable initial response (within 24 hours) to CBZ. Ensuing controlled studies further confirmed the utility of CBZ in initial pain management, and CBZ became a mainstay of TN treatment.

CBZ remains the benchmark first-line treatment for TN due to its robust initial efficacy. However, a systematic review examining the efficacy and safety of CBZ in acute and chronic pain conditions revealed that 40%-66% of patients endured adverse effects. Commonly reported adverse effects of CBZ include somnolence, dizziness, double vision, rash, nausea, headache, vomiting, tremor, ataxia, disturbed sleep, mood changes, lack of concentration, memory loss, and hyponatremia. In rare circumstances, severe adverse effects may be experienced, including myelosuppression, hepatotoxicity, lymphadenopathy, systemic lupus erythematosus, elevated liver enzymes, hematologic dyscrasias, thrombocytopenia, and aplastic anaemia. It is generally recommended that those with medical histories of cardiac, liver, bone marrow, or renal disease undergo regular blood monitoring, as CBZ may be more likely to produce toxic effects in these patients. In addition, the presence of the HLA-B*15:02 allele found almost exclusively in Asian genealogy warrants genetic testing for patients with Asian lineage to determine their potential risk of CBZ-induced Stevens-Johnson syndrome and toxic epidermal necrolysis that may have life-threatening implications.

In the case of CBZ intolerance, oxcarbazepine (OXC), a keto derivative of CBZ, may be trialled, as the mechanism of action parallels carbamazepine; however, OXC has been shown to have fewer side effects, contraindications, and overall better tolerability. Similar to CBZ, common adverse effects include sedation, dizziness, poor concentration, diplopia, nausea, headache, somnolence, ataxia, and thrombocytopenia, typically experienced to a lesser degree compared to CBZ. Of note, the incidence of hyponatremia is dose-dependent and of particular concern, so the use of OXC should be monitored carefully to avoid electrolyte imbalance.

A large retrospective study examining the natural history of classical TN with focus on drug responsiveness and tolerability of CBZ and OXC demonstrated robust initial responsiveness ranging between 98% (CBZ) and 94% (OXC). However, following mean periods of approximately 8.6 (CBZ) and 13 (OXC) months, a significant proportion of patients (27% CBZ and 18% OXC) developed intolerability and required subsequent dosage reduction to inadequate levels for appropriate pain management. CNS disturbances, including somnolence, postural unbalance, and dizziness, were the most prominent causes of treatment discontinuation in patients treated with CBZ, while somnolence, postural unbalance, and hyponatremia were the primary causes for discontinuation of OXC.

In addition, a quantitative examination of the frequency of adverse effects and overall tolerability in patients receiving CBZ and OXC for the treatment management of neuralgiform pain conducted by Besi et al. found that dosage increases sufficient for pain management subsequently increased adverse cognitive effects (i.e., memory and concentration disturbances). More specifically, they found that a standard one-unit dosage increase resulted in a 50% increase in the likelihood of worsening side effects and eventual incapacity to reach therapeutic dosage requirements for adequate pain suppression. Of note, a review by Taylor et al. analyzing the treatment of CBZ for classical TN over a sixteen-year period found a significant drop in efficacy by year four with an overall 44% failure rate, requiring alternative treatment.

Alternatives to CBZ and OXC Gabapentin The efficacy of gabapentin for the treatment of TN has not been clearly demonstrated. However, clinical experience shows better tolerability over CBZ or OXC, albeit with lower efficacy. Gabapentin is still associated with somnolence, dizziness, headache, confusion, nausea, and hyperlipidemia. Nevertheless, gabapentin may be used for patients who are intolerant to or for whom CBZ or OXC are ineffective.

A recent two-year, real-life prospective study by Heinskou et al. aimed at evaluating the prognosis of medically-treated TN in a highly structured multidisciplinary management program. The most frequently utilized drugs at the start of the study were OXC (29%), CBZ (28%), and gabapentin (28%). During the two-year follow-up period, however, 60% of patients experienced a change in the prescribed type or number of medications, and treatment discontinuation occurred in 23% of patients. Although a tightly regulated, individualized drug treatment regimen resulted in a favourable prognosis for nearly half of the patients analyzed at the two-year mark, 45% of patients initially enrolled in the study were lost to follow-up, and a significant number of patients (32%) reported a poor outcome (no pain reduction in 23% or a worsening of pain in 9%). Moreover, a large subset of patients (27%) were referred to surgery due to refractoriness or intolerability, though the optimal time for referral to surgery remains an important unanswered question. The authors do suggest that optimization of treatment "should be done before patients are considered medically refractory".

Despite the favourable tolerability of OXC, a long-term cohort study comparing OXC and surgical management of intractable TN found that effectiveness was short-term, subsequently necessitating surgical intervention as a rescue therapy. Referral to a neurosurgeon varied between 3 months to 11 years following initiation of medical therapy. Surgery was associated with a better outcome than OXC and the authors concluded that patients can benefit substantially from having surgery earlier in the disease process.

In summary, there is a high likelihood (>50%) that, over time, TN patients initially responsive to medical therapy will become medically refractory, failing to respond to alterations in medication type or dosage increases. Ultimately, as outlined above, a consequence of medical therapy is the marked probability of developing intolerance resulting from dosage requirements exceeding safe levels, significantly limiting its use. The long-term efficacy of medical therapy is compromised by intolerability, and over time, intractability of pain.

Surgery has historically been indicated for those who become intolerant or resistant to the ever-increasing dosage requirements required to sustain the efficacy of medical therapy. However, there is no consensus as to the number of failed medical treatments necessary to render a patient appropriate for surgical referral. Despite limited evidence available regarding the optimal time to surgical referral(36), in many patients, pain becomes increasingly intractable with disease duration(31). Therefore, there is a need for further evaluation of the potential benefits of early surgery.

Surgical According to the American Academy of Neurology (AAN) and the European Federation of Neurological Societies (EFNS) guidelines on TN management, when medical therapy becomes ineffective due to poor pain control or intolerability, referral for surgery is the next reasonable step. Below are outlined the three most common surgical approaches to treat TN.

Microvascular Decompression (MVD):

In 1932, neurosurgeon Walter Dandy noted consistent neurovascular compression (NVC) and dorsal root abnormalities in a significant portion of TN patients. Although Dandy's hypothesis was met with criticism, decompressive surgery gained attention as more evidence regarding NVC and the benefit of decompression surfaced. With growing emphasis on NVC as the putative mechanism responsible for TN, Peter Jannetta aimed to refine and legitimize the MVD procedure utilized today. Restorative decompressive surgery (i.e., MVD) is now the preferred surgical treatment in medically refractory classical TN with known NVC.

The purpose of MVD is to mobilize the offending vessel, typically the superior cerebellar artery, away from the root entry zone (REZ) by interposing shredded Teflon at the point of compression to prevent further contact. Although the mechanism of action of MVD is not yet fully understood, decompression may allow for reduced sensitivity and eventual remyelination of the CNV. Remyelination, however, is not an immediate process and it cannot be presumed that remyelination is the cause of immediate pain relief following an MVD; it is plausible that other unknown pathophysiological mechanisms are at play.

Because of its robust efficacy, MVD remains the principal surgical option for medically refractory classical TN in appropriate surgical candidates. Very early reports indicated immediate postoperative pain relief in ~82% of patients directly following surgery and maintained in ~70% of patients at the 10-year mark. A more recent systematic review reported similar immediate postoperative pain relief occurring in 83.5% of patients. Reported rates of pain recurrence are highly variable across studies. A commonly quoted figure is that pain recurrence generally develops within 2 years of surgery in approximately 25% of patients, with a 2-4% annual recurrence rate thereafter.

While MVD is the standard surgical procedure for TN associated with NVC, it is not without the potential risk of complications. Reported complications of MVD include hearing impairment and loss, tinnitus, vertigo, ataxia, diplopia, cerebrospinal fluid (CSF) leak, meningitis, hemifacial paresis, and hypoesthesia. Given the invasive nature of MVD, major complications include the rare but serious risk of cerebral hematoma, supratentorial and brainstem ischemia and infarction, and death. Contraindications to MVD may include comorbidities affecting tolerance to general anesthesia, disorders affecting blood clotting ability, or multiple sclerosis (MS). MVD has been shown to be less effective and carries a high risk of complications for TN secondary to MS, though some neurosurgeons consider it in MS patients with evidence of NVC on imaging. Recent work suggests, however, that NVC may not play a role in the development and maintenance of MS-associated secondary TN.

For patients in whom NVC is not identified at the time of surgery, or in those with idiopathic TN, a variant of MVD called internal neurolysis (IN) may be performed. IN, also referred to as "nerve-combing," is a microsurgical procedure whereby the surgeon uses a blunt-tip instrument to dissect the cisternal portion of the CNV into multiple nerve fascicles. A recent systematic review examining surgical outcomes of IN found that 85%-94.6% of patients had an excellent immediate postoperative outcome, with a 3.9%-17% range of recurrence one-year postoperatively. Given the destructive nature of the procedure, facial numbness is the primary complication of IN, occurring in ~96% of patients. However, facial numbness may likely be transient in a significant portion of patients, decreasing to 1%-10% over time. Additionally, major complications such as corneal ulceration and anesthesia dolorosa have rarely been reported.

Invasive surgical techniques, such as MVD and IN, are certainly highly effective treatment options, providing durable pain relief for a large portion of TN patients. However, the small, but real risk of major and minor complications limits their use to medically fit, typically younger patients, usually with the most severe forms of TN pain and a lengthy history of medical-refractoriness. Accordingly, less-invasive surgical approaches may be appealing to a number of TN patients.

Gamma Knife Stereotactic Radiosurgery (GK-SRS):

Stereotactic radiosurgery (SRS) was developed in 1951 by Swedish neurosurgeon Lars Leksell. The technique uses radioactive cobalt-60 isotope sources to produce converging radiation beams intersecting a target volume, and was ultimately adapted for treating TN. Regarded as the least invasive neurosurgical approach, GK-SRS is entirely non-invasive other than the use of stereotactic headframe immobilization. In a single session, GK-SRS delivers a highly concentrated dose of ionizing radiation to a precise treatment target along the CNV (see below). GK-SRS targets the CNV with high precision and accuracy, and the distribution of the therapeutic radiation dose is precisely tailored to treatment margins so that irradiation of surrounding normal healthy tissues beyond treatment margins is minimal.

The optimal GK-SRS target in TN is controversial. However, two target zones are most frequently used: dorsal root entry zone (DREZ) (anterior to the junction of the CNV with the pons) and the retrogasserian zone (RGZ) (posterior to the Gasserion ganglion and anterior to the DREZ), also referred to as the mid-cisternal segment. Comparative and retrospective studies have shown more favourable outcomes in the RGZ approach due to a shorter time to pain relief, higher likelihood of complete pain relief without medication, a lower incidence of bothersome facial numbness, and a lower rate of dry eye syndrome. Additionally, the ideal radiation prescription dose has not yet been clearly defined. However, in most available literature, maximal doses range from 70-90 Gy; it is thought that dosing which is too low renders the procedure ineffective for long-term pain control, while too high a dose results in post-procedural complications (e.g., facial paresthesias). Thus, finding a balance between 70-90 Gy may be optimal; indeed, Lee et al. found that administering a mean dose of 80 Gy yielded earlier and more durable postoperative pain relief.

GK-SRS offers a minimally invasive treatment alternative for patients who are refractory to medical or other surgical treatment, are not candidates for a more invasive procedure requiring general anesthesia, or those with coagulation disorders or taking medications affect clotting factors and anticoagulant proteins. GK-SRS, however, may be less suitable for patients in whom rapid pain relief is critical, as pain relief is generally gradual (8-12 weeks).

There is evidence to support long-term safety and efficacy of GK-SRS for the treatment of TN. One such study reported in Radiosurgery (2006) demonstrated the durability of primary GK-SRS for extended pain control. The authors found that half of the 87% of patients who achieve complete pain control remain pain-free for approximately six years, with a low incidence of side effects (5%). These findings support other reports on the benefit of primary GK-SRS in patients without any prior neurosurgical intervention for TN. For example, Pollock et al. found a 3-year complete pain-free actuarial rate of 49% in patients with previous surgical procedures, compared to 55% in patients where GK-SRS was their primary treatment.

Similarly, Huang et al. assessed the outcome of primary and repeat GK-SRS for the treatment of idiopathic TN and concluded that actuarial response rate (66% at 3 years) was similar to that of other research evaluating GK-SRS as a primary treatment, with half of the patients experiencing pain freedom without the use of medication over a mean follow-up period of 5.7 years. Caveats to these findings include the lack of randomization leading to potential selection bias. Nevertheless, these findings demonstrate that primary GK-SRS may provide durable pain control and establishes the foundation for eliciting further controlled studies.

Pooled data gathered by Tuleasca et al. in their systematic review and meta-analysis of GK-SRS for TN provides the strongest evidence to date supporting GK-SRS as a safe and effective therapy for refractory TN. Forty-five GKS SRS studies (5687 patients) were analyzed based on freedom from pain (FFP), time to pain relief (TTPR), recurrence rates, time to recurrence, and presence of hypesthesia or other complications and their respective time points. Mean FFP outcome with or without medication adjustment was 84.8% and mean FFP outcome without the need for medication entirely was 53.1%, with TTPR ranging from 15-78 days. Mean pain recurrence rate was 24.6%, occurring between 7.5-20.4 months. Additionally, the maintenance of pain relief at 7 and 10 years was noteworthy in five studies, ranging between 22% and 59.7% (7 years) and 30% and 45.3% (10 years). Incidence of facial sensory dysfunction (i.e., hypesthesia) is the most significant complication of GK-SRS (21.7%), occurring between 6 to 36 months. However, the development of bothersome or very bothersome hypesthesia occurred in only a small proportion of patients (0%-17.3% mean = 3.1%). Other rare side effects included dry eye, deafferentation pain, and keratitis. In 27/45 GK-SRS studies, there were no reported side effects at all. In addition, post GK-SRS associated malignancies are rare, with a cumulative incidence of 0.00045% over 10 years. Other uncommon complications include dry eye (1.9%-22.4%) and keratitis (2.7%-7%).

Although there is substantial evidence in support of GK-SRS for the treatment of medically refractory TN, there remains a notable gap in the literature exploring very early GK-SRS. Of particular importance, of the 45 studies reviewed by Tuleasca et al., only one retrospective study analyzed GK-SRS when used exclusively as the primary surgical treatment in TN. Mousavi et al. reported initial pain relief in 88% of patients, ranging from three days to six months after treatment. The authors found that earlier GK-SRS treatment (within 3 years of pain onset) resulted in earlier pain relief (median of 1 week) compared to 6 weeks for patients whose pain had been present longer than three years prior to GK-SRS. Additionally, a longer duration of adequate pain control was seen in a larger percentage of patients whose pain history was 3 years or less (1 year 93%, 10 years 73%) compared to those whose pain persisted longer prior to GK-SRS treatment (1 year 63%, 10 years 28%). Moreover, a longer interval of pain relief without medication (89% at 3 years) was seen in a greater proportion of patients with a history of pain <3 years compared to those with >3-year history of pain (52% at 3 years). Patients with a history of pain for >3 years prior to GK-SRS had an 8% likelihood of being pain-free without medication by year 5 and 0% at year 10, compared to 73% and 40%, respectively in patients with pain <3 years.

Furthermore, a recent international multicenter study proposed consideration of earlier radiosurgery (within 4 years of diagnosis), as they found that patients had a shorter interval to pain relief and yielded significant decreases in adjunct medication utilization within this time-frame. Taken together, these findings point to the potential value of early GK-SRS treatment in providing faster and more durable medication-free pain relief, with a very low rate of adverse side effects.

Rationale Despite the high likelihood of experiencing adverse effects and very low-quality evidence supporting its use before offering surgery, there is a strong recommendation that CBZ be implemented as the standard of care treatment for TN. While the initial efficacy of medical therapy argues for implementing pharmaceutical treatment as the first line approach, long-term efficacy is hindered by a high likelihood of developing intolerance to treatment. However, no definitive data is currently available to determine how many trials of medication are required before referral to surgery, nor has an optimal time for surgical referral been established. Although some guidelines state that up to three groups of medications be trialed, some experts believe that patients who fail first-line medical therapy are unlikely to respond to other medications and should be referred for surgery earlier.

Ultimately, it remains the responsibility of the treating clinician to determine when a patient should be considered for surgical intervention. However, care pathways for TN patients are extremely variable due to the wide range of specialists consulted and inconclusive treatment recommendations available. There is evidence, however, that patients refractory to medical therapy prefer earlier surgery.

As surgical intervention is implicated in a significant percentage of patients (>50%) who ultimately become medically refractory, variability in treatment recommendations and subsequent delay in surgical referral may impede access to treatment prior to the critical period in which acute pain transitions to more chronic, difficult-to-treat pain. Pain chronification results from the extended imbalance of pain amplification and inhibition, both peripherally and centrally, leading to neuronal hyperexcitability and increased pain hypersensitivity to innocuous stimuli. Consequently, increasing evidence indicates distinct structural and functional maladaptive remodelling of the central and peripheral nervous system of individuals with chronic pain disorders. Certainly, an argument can therefore be made that earlier surgical intervention prior to pain chronification has a sound theoretical rationale.

While MVD is generally the initial surgical treatment recommendation for classical TN patients, it is not without its risk of serious complications and may not be appropriate be in patients unfit for open craniotomy or those diagnosed with secondary or idiopathic TN. Similarly, percutaneous procedures also carry at least some risk of catastrophic complications, do require either general anesthesia or conscious sedation, and are associated with a relatively high recurrence rate over time. GK-SRS, however, is well-tolerated, and its long-term safety and efficacy are well-established. Reported complications are typically transient, and severe, permanent complications are exceedingly rare.

Current recommendations state that surgical complications ought to be balanced against the adverse effects of long-term medical therapy when determining an appropriate course of treatment. Accordingly, it is pertinent to consider that the number needed to harm (NNH) for the most significant complication of GK-SRS (i.e., hypesthesia) is approximately 4.7 compared to approximately 2.6 for at least one adverse effect of CBZ.

Limitations and gaps in the current literature examining primary GK-SRS for the treatment of TN have motivated the objective of this research. Whilst some of the literature discussed here indicates that earlier treatment with GK-SRS results in durable long-term pain remission, this research has not yet been evaluated in a controlled clinical trial. Thus, there is a need for such controlled research to provide further evidence in support of the safety and efficacy of GK-SRS as a primary intervention for TN and to guide future treatment recommendations.

If GK-SRS, implemented as a first-line treatment for TN, proves safe and effective, then this research would represent a paradigm shift in TN management. Clinically, these findings will translate to less ambiguity in optimal time to surgical referral and an increased willingness to refer patients for earlier surgery. As a result, TN treatment guidelines may adopt firmer recommendations for earlier surgical treatment, enabling both clinicians and patients with more informed decision-making potential. Validating the evidence in favour of GK-SRS as a viable first-line treatment option may mitigate potentially detrimental repercussions of prolonged disease duration on pain chronification and overall detriment to quality of life with extended insufficient medical management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of classical or idiopathic TN, based on clinical history and MRI scan
* Onset of pain within 2 years prior to enrolment
* Not deemed medically refractory (defined as uncontrolled pain despite ≥2 medication trials, not requiring escalating dose)
* If currently on medication, on stable dose x at least 3 months

Exclusion Criteria:

* Secondary TN
* Bilateral TN
* Any contraindications to undergoing GK-SRS
* Any prior cranial radiation
* Any prior surgical intervention for TN
* History of psychiatric diagnoses within 2 years of study participation, or uncontrolled, concurrent psychiatric illness (e.g., depression with recent suicide attempts)
* Females who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure--pain | 2 years after the day of GK-SRS treatment, for participants in the Experimental Arm. 2 years after enrolment, for participants in the No-intervention Arm.
  The primary endpoint is satisfactory pain control at 2 years after GK-SRS treatment (for Experimental Arm) or 2 years after enrolment in the Non-intervention Arm, measured using Barrow Neurological Institute Facial Pain Scale (BNI). Satisfactory pain control = BNI I, II, IIIa
  Barrow Neurological Institute Facial Pain Scale (BNI) I - no pain, no medication II - occasional pain, no medication required III - some pain, adequately controlled with medication IIIa - no pain, continued medication IIIb - persistent pain, controlled with medication IV - some pain, not adequately controlled with medications V - severe pain or no pain relief
  (lower scores indicate better outcome)

SECONDARY OUTCOMES:
Secondary outcome measure - treatment-related adverse events | At 6, 12, 24 months, and 5 years after the day of GK-SRS treatment, for participants in the Experimental Arm. At 6, 12, 24 months, and 5 years after enrolment, for participants in the No-intervention Arm
  Worst incidence of treatment-related adverse events by treatment arm. Adverse events will be determined using the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Secondary outcome measure - medication | Experimental Arm: Baseline visit; GK-SRS treatment visit; follow-up visits 6, 12, 24 months, and 5 years after day of GK-SRS treatment. No-intervention Arm: Baseline visit; follow-up visits 6, 12, 24 months, and 5 years after enrolment
  Pain medication equivalent dose measured with the Medication Quantification Scale version III
  (lower scores indicate better outcome)
Secondary outcome measure - complete pain relief | 2 years after the day of GK-SRS treatment
  Score of 'BNI I' on the Barrow Neurological Institute Facial Pain Scale (BNI)
  Barrow Neurological Institute Facial Pain Scale (BNI) I - no pain, no medication II - occasional pain, no medication required III - some pain, adequately controlled with medication IIIa - no pain, continued medication IIIb - persistent pain, controlled with medication IV - some pain, not adequately controlled with medications V - severe pain or no pain relief
  (lower BNI score indicates better outcome)
Secondary Outcome Measure - long term satisfactory pain relief | 5 years after day of GK-SRS treatment
  Proportion of patients with satisfactory pain control at 5 years after Gamma Knife treatment, measured using Barrow Neurological Institute Facial Pain Scale (BNI).
  Satisfactory pain control = BNI I, II, IIIa Barrow Neurological Institute Facial Pain Scale (BNI) I - no pain, no medication II - occasional pain, no medication required III - some pain, adequately controlled with medication IIIa - no pain, continued medication IIIb - persistent pain, controlled with medication IV - some pain, not adequately controlled with medications V - severe pain or no pain relief (lower scores indicate better outcome)
Secondary Outcome Measure - facial numbness | At 6, 12, 24 months, and 5 years after GK-SRS treatment
  Presence and severity of facial numbness in the Experimental Arm after GK-SRS treatment.
  Measured using the Barrow Neurological Institute Facial Numbness Scale (BNI) I= no facial numbness II= mild facial numbness that is not bothersome III= somewhat bothersome facial numbness IV= very bothersome facial numbness
Secondary outcome measure - crossover | At 6, 12, 24 months, and 5 years after enrolment
  Number of patients crossing over from medication arm (i.e., No-intervention arm) to surgery during follow up period
Secondary outcome measure - repeat surgical referral | At 6, 12, 24 months, and 5 years after GK-SRS treatment
  Number of patients in GK SRS arm referred for repeat surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lussoso A, Patel S, Hussain W, Knash M, Bowden G, Wheatley M, Vu NK, Sankar T. Ultra-early Gamma Knife stereotactic radiosurgery for trigeminal neuralgia (URGEnt-TN): study protocol for a single-center, two-arm, parallel group design, pragmatic, noninferiority, phase II, randomized controlled trial with intention-to-treat analysis for pre-refractory GK-SRS in classical or idiopathic TN. Trials. 2025 Dec 4;27(1):15. doi: 10.1186/s13063-025-09321-8. PMID 41345955